CLINICAL TRIAL: NCT04918394
Title: Assessment of Mold Exposure in Asthmatic Children Follow-up in Nord and Pas-De-Calais Departments, France, and Impact on Asthma Control
Brief Title: Mold Exposure and Impact on Asthma Control in French Asthmatic Children
Acronym: CHAMPIASTHMA
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_49; 2019-A03310-57 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Asthma in Children
Keywords: Asthma; Children; Mold; Moisture; Asthma Control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma patients unexposed to mold / moisture: No mold / moisture exposure is defined by a negative response to all of the 5 following questions, asked in the form of a parent-completed declarative questionnaire regarding the child's primary living home.
  Interventions: Other: Questionnaire of Mold / moisture exposure
- Asthma patients exposed to mold / moisture: Mold / moisture exposure is defined by a positive response to at least one of the 5 following questions, asked in the form of a parent-completed declarative questionnaire regarding the child's primary living home.
  Interventions: Other: Questionnaire of Mold / moisture exposure

INTERVENTIONS:
Other: Questionnaire of Mold / moisture exposure — Mold / moisture exposure is assessed by the 5 following questions, whose positive response has been associated with the actual presence of mold in the household (according to data from the literature data), asked in the form of a parent-completed declarative questionnaire regarding the child's primary living home:
  * Presence of visible mold
  * Impression of dampness
  * Apparent dampness
  * Existence of recent water damage in the last year
  * Presence of a moldy odor

SUMMARY:
Observational, multicenter, study conducted in 12 hospitals in the Nord and Pas-De-Calais departments. The aim of this study is to describe the relationship between reported exposure to molds and asthma control in a pediatric population.

Each patient followed by a specialized asthma pediatrician in one of the study center will be proposed to participate in the study.

Children aged 1 to < 18 years, with asthma diagnosis, based on the assessment of a specialized physician after a follow-up of at least 6 months Inclusion, non-inclusion and exclusion criteria will be verified by the investigators. The questionnaires will be completed during the consultation, collected by the physician in charge of the consultation and sent to the principal investigator for data entry.

Inclusion will take place over a period of 12 consecutive months from the date of obtaining regulatory approval.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to < 18 years, with asthma diagnosis, based on the assessment of a specialized physician after a follow-up of at least 6 months, Follow-up in one of the study center in Nord and Pas de Calais departments (Lille, Lens, Tourcoing, Valenciennes, Arras, Roubaix, Seclin, Armentières, Calais, Boulogne/mer, Dunkerque, GHICL-Saint Vincent) over an inclusion period of 12 months

Exclusion Criteria:

* Children living ≤ 50% of the weekly time in their primary home (e.g., shared custody)
* Children whose living arrangement characteristics are difficult to analyze (e.g., child accompanied by grandparents or by the parent without primary custody)
* Children whose residence has recently changed, making it impossible to assess the impact of the living arrangement over the past year
* Children living outside of the Nord and Pas-de-Calais departments
* Children whose parents are unable to complete the questionnaire

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children follow-up by a specialized asthma pediatrician in secondary (general hospital) and tertiary care (Lille university hospital) centers.
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Asthma control according to GINA guidelines | At the time of inclusion
  The Global Initiative for Asthma (GINA)guidelines:
  Well controlled Partly controlled Uncontrolled

SECONDARY OUTCOMES:
Asthma control according to Asthma Control Test (ACT) score in children aged 12 years and older: Controlled if ACT ≥ 20 | At the time of inclusion
  Asthma Control Test: Each question is assigned a score between 1 and 5 (the score for the first answer proposal is 1, the second is 2, and so on). The score of the 5 questions is added up to a total score that can vary between 5 and 25. The higher the total score, the better the asthma is controlled.
Asthma control according to pACT score in children aged 1 to 11 years old: Controlled if ACT ≥ 20 | At the time of inclusion
Asthma treatment step according to GINA guidelines: Step 1 to step 4 in children aged < 6 years Step 1 to step 5 in children aged ≥ 6 years | At the time of inclusion
Inhaled corticosteroid doses in µg/day of fluticasone | At the time of inclusion
Acute asthma events in the past 12 months | At the time of inclusion
  Acute asthma events: emergency room visits, hospitalization, general corticosteroid course
Exposure to other indoor pollutants: cigarette smoke (declarative smoking by at least one of the parents) | At the time of inclusion
Exposure to indoor allergens: declarative exposure to animal danders | At the time of inclusion
Exposure to indoor allergens: declarative exposure to house dust mite (carpet, mattress) | At the time of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DESCHILDRE, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (10):
- France (10):
  - Ch Armentieres, Armentières
  - Ch Boulogne-Sur-Me, Boulogne-sur-Mer
  - Ch Calais, Calais
  - CH Dunkerque, Dunkirk
  - Centre Hospitalier de Lens, Lens
  - Hop Jeanne de Flandre Chu Lille, Lille
  - Centre Hospitalier St Vincent, Lille
  - Centre hospitalier de Roubaix, Roubaix
  - Centre Hospitalier de Seclin, Seclin
  - Centre Hospitalier,, Valenciennes

REFERENCES:
- [Derived] Sauvere M, Lejeune S, Chagnon F, Drumez E, Cisterne C, Mordacq C, Thumerelle C, Scalbert M, Le Mee A, Amani M, El Mourad S, Enchery S, Pouessel G, Roussel J, Dartus M, Behal H, Deschildre A. Home exposure to moisture and mold is associated with poorer asthma control in children: CHAMPIASTHMA study. J Allergy Clin Immunol Glob. 2025 Jan 17;4(2):100415. doi: 10.1016/j.jacig.2025.100415. eCollection 2025 May. PMID 40130077